CLINICAL TRIAL: NCT03024866
Title: A Multi-Center Retrospective-Prospective Matched Pairs Cohort Study to Assess Long-term Clinical Outcomes of Non-melanoma Skin Cancer Patients Treated With eBx Compared to Non-melanoma Skin Cancer Patients Treated With Mohs Surgery
Brief Title: Comparison of eBX and Mohs Surgery for Treatment of Early-stage Non-melanoma Skin Cancer a Matched Pair Cohort Study.
Status: Completed | Type: Observational
Sponsor: Xoft, Inc. (Industry)
Collaborators: Eminence Clinical Research, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CTPR-0014
Record Dates: First submitted 2017-01-11; First posted 2017-01-19 (Estimated); Results first posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Nonmelanoma Skin Cancer
MeSH Terms: interventions — Mohs Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Electronic Brachytherapy: Procedure/Surgery: Electronic Brachytherapy:
  Previously completed treatment for non-melanoma skin cancer using Xoft eBx Electronic Brachytherapy System. High-dose-rate electronic brachytherapy (EBT) provides a non-surgical treatment option for non-melanoma skin cancer (NMSC).
  Interventions: Procedure: Electronic Brachytherapy
- Mohs Surgery: Previously completed treatment for non-melanoma skin cancer using Mohs Surgery:
  Uniquely orients, maps, and processes removed tissue, permitting the microscopic evaluation of virtually 100% of the specimen margins. The completeness of this margin control permits the accurate identification and removal of all tumor extensions under the microscope. Tissues in Mohs surgery are processed as modified frozen sections which allow the accurate and rapid interpretation of most skin cancers.
  Interventions: Procedure: Electronic Brachytherapy

INTERVENTIONS:
Procedure: Electronic Brachytherapy — A group receives High-dose-rate electronic brachytherapy (EBT) which provides a non-surgical treatment option and the other group receives Mohs surgery. This matched-pair cohort study compared the outcomes of treatment with EBT to those of Mohs surgery in patients with NMSC.
  Other Names: Mohs Surgery

SUMMARY:
This is a retrospective-prospective study design. Patients who completed treatment approximately 3 years (range of 2-4 years) at time of IRB approval of this study will be identified and any existing data in the patient's record will be collected in addition to conducting office visits for long-term follow-up.

DETAILED DESCRIPTION:
This is a retrospective-prospective study design. Patients who completed treatment approximately 3 years (range of 2-4 years) at time of IRB approval of this study will be identified and any existing data in the patient's record will be collected in addition to conducting office visits for long-term follow-up. The study will include 2 parts:

1. Retrospective chart review: Collect data from patient records who completed treatment a minimum of 2 years prior to study onset and determine the feasibility of doing a matched pair cohort study comparison of eBx versus Mohs surgery. The history, demographic and treatment data will be retrospectively collected from up to 320 subjects previously treated with eBx for the treatment of NMSC and up to 320 subjects previously treated with Mohs surgery for the treatment of NMSC.
2. Prospective Follow-up: Patients will return for long-term follow-up visits for the investigators to assess the lesion site, document absence of recurrence/ absence of recurrence, toxicities, and collect patient reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Previously completed treatment for non-melanoma skin cancer using Xoft eBx Electronic Brachytherapy System or Mohs surgery;
2. Provides informed Consent;
3. Greater than 40 years of age;
4. Pathological diagnosis confirmed to be squamous cell or basal cell carcinoma prior to treatment;
5. Cancer Staging included in this study:

   * Stage 0: Tis, N0, M0
   * Stage 1: T1, N0, M0
   * Stage 2: T2, N0, M0 and ≤ 4cm in diameter

Exclusion Criteria:

1. Target area is adjacent to a burn scar
2. Any prior definitive surgical resection of the cancer, prior to Radiation Treatment
3. Known perineural invasion
4. Actinic Keratosis
5. Known spread to regional lymph nodes
6. Known metastatic disease

Min Age: 41 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 320 subjects treated with eBx and up to 320 subjects treated with Mohs surgery will have data collected retrospectively from the patient's medical records, and prospectively at the time of the follow-up visit for those who agree to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 369 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Patel, MD, Principal Investigator — Good Samaritan Radiation Oncology; Robert Strimling, Principal Investigator — Strimling Dermatology, Laser, and Vein Institute
Locations (4):
- United States (4):
  - Kenneth A. Miller, PC, Los Gatos, California
  - Dermatology & Laser Center of San Diego, San Diego, California
  - Dermatology and Laser Center of San Diego, San Diego, California
  - Strimling Laser and Vein Institute, Las Vegas, Nevada

REFERENCES:
- [Result] Patel R, Strimling R, Doggett S, Willoughby M, Miller K, Dardick L, Mafong E. Comparison of electronic brachytherapy and Mohs micrographic surgery for the treatment of early-stage non-melanoma skin cancer: a matched pair cohort study. J Contemp Brachytherapy. 2017 Aug;9(4):338-344. doi: 10.5114/jcb.2017.68480. Epub 2017 Jun 23. PMID 28951753

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Identify and collect any existing data from the patients record and conduct office visits on patients with non-melanoma skin cancer who underwent treatment with either eBx or Mohs and completed treatment approximately 3 yrs prior (range of 2-4 years) to asses long-term outcomes of treated areas.
Pre-assignment Details: N/A This is a retrospective-prospective study design.
Groups:
- Mohs Surgery: Previously completed treatment for non-melanoma skin cancer using Mohs Surgery
- Electronic Brachytherapy: Previously completed treatment for non-melanoma skin cancer using Xoft eBx Electronic Brachytherapy System
Period: Overall Study
Arm/Group | Mohs Surgery | Electronic Brachytherapy
Started | 181 (Patient's return for follow-up visit to asses long-term outcomes of previous treatment with Mohs.) | 188 (Patient's return for follow-up visit to asses long-term outcomes of previous treatment with eBx.)
Completed Enrollment | 181 | 188
Completed | 181 | 188
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Units Other Than Participants: Lesions Analyzed
Groups:
- Electronic Brachytherapy: Previously completed treatment of 1 or more non-melanoma skin cancer lesions per participant using Xoft eBx Electronic Brachytherapy System
- Mohs Surgery: Previously completed treatment of 1 or more lesions per participant for non-melanoma skin cancer using Mohs Surgery
- Total: Total of all reporting groups
Arm/Group | Electronic Brachytherapy | Mohs Surgery | Total
Number analyzed (Participants) | 188 | 181 | 369
Number analyzed (Lesions Analyzed) | 208 | 208 | 416
Age, Customized [Mean (Standard Deviation); unit: years]
  eBx | 80.8 (7.2) | 76.6 (8.8) | 78.7 (8.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 65 | 61 | 126
  Male | 123 | 120 | 243
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 0 | 1 | 1
  Caucasian Non-Hispanic | 186 | 180 | 366
  Asian Pacific Islander | 2 | 0 | 2
Lesions by Size [Number; unit: lesions] — 0 ≤1cm 0 >1cm and ≤2cm 0 >2cm and >2cm 0 N/A
  lesions
    Lesions less than 1cm | 57 | 57 | 114
    Lesions greater than 1cm less than 2cm | 146 | 146 | 292
    Lesions greater than 2cm less than 3cm | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Absence of Local Recurrence at Treatment Site(s) Greater or Equal to 3 Years Follow-up
Description: Subjects treated with Xoft eBx or MMS over 3 years prior were called in for a long-term prospective visit, consented, and assessed for skin cancer recurrence at the previously treated site.
Time Frame: Range greater or equal to 3 years post last Xoft eBx or MMS treatment at the time of study start at1 long-term prospective visit by study completion.
Measure: Number; unit: participants
Units Other Than Participants: Lesions Analyzed
Groups:
- Electronic Brachytherapy: Previously completed treatment of 1 or more lesions per participant for non-melanoma skin cancer using Xoft eBx Electronic Brachytherapy System
  Electronic Brachytherapy: High-dose-rate electronic brachytherapy (EBT) provides a non-surgical treatment option for non-melanoma skin cancer (NMSC). This matched-pair cohort study compared the outcomes of treatment with EBT to those of Mohs surgery in patients with NMSC.
- Mohs Surgery: Previously completed treatment of 1 or more lesions per participant for non-melanoma skin cancer using Mohs Surgery
  Electronic Brachytherapy: High-dose-rate electronic brachytherapy (EBT) provides a non-surgical treatment option for non-melanoma skin cancer (NMSC). This matched-pair cohort study compared the outcomes of treatment with EBT to those of Mohs surgery in patients with NMSC.
Arm/Group | Electronic Brachytherapy | Mohs Surgery
Number analyzed (Participants) | 188 | 181
Number analyzed (Lesions Analyzed) | 208 | 208
participants
  Participants Analyzed | 188 | 181
  Absence of Local Recurrence | 187 | 181
  Lesions Analyzed | 208 | 208

2. Secondary Outcome: Comparison of Late Toxicities Related to eBx vs. Mohs Treatment Using A Chronic Toxicity Questionnaire Based on Physician Assessment at Long-term Prospective Visit
Description: Subjects treated with Xoft eBx or MMS over 3 years prior were called in for a long-term prospective visit, consented, and assessed to determine if late toxicities occurred at the previously treated site with Xoft eBx or MMS.
Time Frame: as for outcome 1
Measure: Number; unit: lesions
Units Other Than Participants: Lesions Analyzed
Groups:
- Electronic Brachytherapy; Mohs Surgery: Previously completed treatment of 1 or more lesions per participant for non-melanoma skin cancer
Arm/Group | Electronic Brachytherapy | Mohs Surgery
Number analyzed (Participants) | 188 | 181
Number analyzed (Lesions Analyzed) | 208 | 208
lesions | 138 | 143

3. Secondary Outcome: Comparison of Long-term Cosmetic Outcomes for Lesions Treated for NMSC With eBx vs. Mohs
Description: Subjects treated with Xoft eBx or MMS over 3 years prior were called in for a long-term prospective visit, consented, and an assessment of cosmetic outcome occurred at the previously treated site with Xoft eBx or MMS.
Time Frame: as for outcome 1
Measure: Number; unit: lesions
Units Other Than Participants: Lesions Analyzed
Arm/Group | Electronic Brachytherapy | Mohs Surgery
Number analyzed (Participants) | 188 | 181
Number analyzed (Lesions Analyzed) | 208 | 208
lesions | 203 | 199

4. Secondary Outcome: Chronic Toxicities
Description: Subjects treated with Xoft eBx or MMS over 3 years prior were called in for a long-term prospective visit, consented, and assessed to determine if there were any chronic toxicities found at the previously treated site with Xoft eBx or MMS.
Time Frame: as for outcome 1
Population: Analysis same as late toxicities.
Measure: Count of Units; unit: Lesions Analyzed
Units Other Than Participants: Lesions Analyzed
Arm/Group | Electronic Brachytherapy | Mohs Surgery
Number analyzed (Participants) | 188 | 181
Number analyzed (Lesions Analyzed) | 208 | 208
Lesions Analyzed | 138 | 143

5. Secondary Outcome: Patient Survey for Reporting Patient Reported Outcomes (PRO)
Description: Subjects treated with Xoft eBx or MMS over 3 years prior were called in for a long-term prospective visit, consented, then subjects completed a Patient Satisfaction Score: min=0, max=60, with 60 as the maximum positive or favorable response.
Time Frame: Range greater or equal to 3 years post last Xoft eBx or MMS treatment at the time of study start, with 1 long-term prospective visit by study completion.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Electronic Brachytherapy | Mohs Surgery
Number analyzed (Participants) | 188 | 181
score on a scale | 54.0 (9.0) | 56.0 (5.3)

ADVERSE EVENTS:
Time Frame: Patients have been followed for 2.6 to 4.3 years after EBT, and 2.3 to 5 years following MMS.
Description: All additional adverse events that were collected have been reported. The only adverse events reported were all skin toxicities from CTCAE.
Arm/Group | Mohs Surgery | Electronic Brachytherapy
All-Cause Mortality (participants affected / at risk) | 0/181 | 0/188
Serious Adverse Events (participants affected / at risk) | 0/181 | 0/188
Other Adverse Events (participants affected / at risk) | 79/181 | 107/188
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mohs Surgery (N=181) | Electronic Brachytherapy (N=188)
Late toxicities (Skin and subcutaneous tissue disorders) | 79 (181) | 107 (188) — hypopigmentation, hyperpigmentation, erythematous car, telangiectasia, hair loss, fibrosis, atrophy, loss of subcutaneous tissue, hypertrophy/keloid, poor healing/ulceration/erosion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-07): https://cdn.clinicaltrials.gov/large-docs/66/NCT03024866/Prot_SAP_000.pdf